CLINICAL TRIAL: NCT02458690
Title: eIMPACT Trial: Modernized Collaborative Care to Reduce the Excess CVD Risk of Older Depressed Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jesse Stewart, Professor of Psychology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1411802537; R01HL122245 (NIH)
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Depression; Major Depressive Disorder; Dysthymic Disorder; Depressive Symptoms; Cardiovascular Diseases; Heart Diseases; Coronary Artery Disease; Stroke
Keywords: Primary Care; Older Adults; Computerized and Telephonic Psychotherapy; Cognitive-Behavioral Therapy; Antidepressant Medications
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Dysthymic Disorder; Cardiovascular Diseases; Heart Diseases; Coronary Artery Disease; Stroke | interventions — Cognitive Behavioral Therapy; Primary Health Care; Selective Serotonin Reuptake Inhibitors; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- eIMPACT (Experimental): eIMPACT is a 12-month, modernized, collaborative, stepped care intervention consisting of (1) computerized and telephonic cognitive-behavioral therapy for depression and (2) select antidepressant medications included in an algorithm optimized for cardiovascular disease risk reduction. It is a collaborative care intervention in which a multidisciplinary team delivers established depression treatments consistent with patient preference. It uses a stepped, flexible, treat-to-target approach that modernizes the IMPACT intervention by harnessing technology to minimize staff and space requirements. Interventions are Beating the Blues, Problem Solving Treatment in Primary Care, and select FDA-approved antidepressants. The treatment team consists of a depression clinical specialist, a supervising MD with expertise in primary care and IMPACT, and the patients' primary care providers.
  Interventions: Behavioral: Beating the Blues (BtB); Behavioral: Problem Solving Treatment in Primary Care (PST-PC); Drug: Antidepressant Medications
- Usual Care (Active Comparator): Patients and their primary care providers are informed of the depressive disorder diagnosis, and follow-up is encouraged. There are no restrictions on the care received. The Eskenazi Health primary care clinics utilize a team care approach, with PCPs supported by embedded behavioral health clinicians and affiliated psychiatrists.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Beating the Blues (BtB) — BTB is a widely used, empirically supported, stand-alone CBT program for depression designed for primary care patients and appropriate for adults with little computer experience and a 5th-6th grade reading level. BtB utilizes an interactive, multimedia format to deliver eight 50-minute, weekly therapy sessions. Although sessions are tailored to each patient's problems, general topics include challenging dysfunctional thoughts, activity scheduling, problem solving, graded exposure, task breakdown, sleep management, and relapse prevention. Patients are also assigned tailored homeworks that are customized to their needs and reviewed at the start of each session.
  Other Names: Cognitive-Behavioral Therapy (CBT); Computer-Based Psychotherapy
  Arms: eIMPACT
Behavioral: Problem Solving Treatment in Primary Care (PST-PC) — PST-PC is a manualized, empirically supported CBT developed for use by healthcare professionals in primary care. The focus of the 6-10 30-minute sessions is teaching patients approaches for solving current problems contributing to depression. We are delivering PST-PC via telephone.
  Other Names: Cognitive-Behavioral Therapy (CBT); Telephonic Psychotherapy
  Arms: eIMPACT
Drug: Antidepressant Medications — The IMPACT treatment manual provides guidelines for using antidepressants, such as selecting a medication, titrating, switching to another medication, managing side effects, and avoiding drug interactions. To optimize eIMPACT for CVD risk reduction, we have restricted the IMPACT list of antidepressants to SSRIs (sertraline, escitalopram, paroxetine, fluoxetine, citalopram), duloxetine, bupropion, and mirtazapine. These medications are FDA approved for the treatment of depression and are the safest from a cardiovascular perspective.
  Other Names: Selective Serotonin Reuptake Inhibitors (SSRIs); Serotonin-Norepinephrine Reuptake Inhibitor (SNRI); Norepinephrine-Dopamine Reuptake Inhibitor (NDRI); Tetracyclic Antidepressant (TeCA)
  Arms: eIMPACT
Other: Usual Care — Patients randomized to usual primary care for depression are informed of their depression diagnosis, encouraged to follow-up with their Eskenazi Health primary care provider, and provided a list of local mental health services. The patient's primary care provider will receive a letter indicating that their patient has a depressive disorder and was randomized to usual care. This letter also provides a list of local mental health services. Like those in the intervention group, usual care patients continue to have access to services that are part of usual care in the targeted systems. There are no restrictions on the care received. The Eskenazi Health primary care clinics utilize a team care approach, with PCPs supported by embedded behavioral health clinicians and affiliated psychiatrists.
  Other Names: Treatment As Usual (TAU)
  Arms: Usual Care

SUMMARY:
The objective of this randomized controlled trial is to evaluate whether the investigators modernized IMPACT intervention for depression (eIMPACT), delivered before the onset of cardiovascular disease (CVD), reduces the risk of future CVD. Participants will be primary care patients who are depressed but do not have a history of CVD. Half of the participants will receive standard depression treatment in primary care (usual care), and the other half will receive one year of eIMPACT, a collaborative stepped care program including antidepressants and computerized and telephonic cognitive-behavioral therapy. To evaluate change in CVD risk, the investigators will measure artery function using ultrasound before and after the 1-year treatment period. It is hypothesized that patients who receive the eIMPACT intervention will have greater improvements in artery function than patients who receive usual care.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the number one killer of American men and women, and its economic burden is substantial and on the rise. Adults with depression are at elevated risk of CVD events and poor CVD prognosis. Unfortunately, past trials of depression treatments have not observed the anticipated cardiovascular benefits. A novel explanation for these null results is that the interventions in these trials, which all involved patients with preexisting CVD, were delivered too late in the natural history of CVD. To begin to evaluate our hypothesis that treating depression before clinical CVD onset could reduce CVD risk, the investigators are conducting a phase II randomized controlled trial of 216 primary care patients aged ≥ 50 years with a depressive disorder and CVD risk factors but no clinical CVD. Patients will be randomized to one year of eIMPACT, our modernized IMPACT intervention, or usual primary care for depression. eIMPACT is a collaborative stepped care intervention involving a multidisciplinary team delivering evidenced-based depression treatments consistent with patient preference. The investigator shave modernized our intervention by incorporating computerized cognitive-behavioral therapy and delivering other treatment components via telephone. Our central hypothesis is that eIMPACT will improve endothelial dysfunction, which is considered a barometer of CVD risk, in depressed adults by decreasing depressive symptoms, autonomic dysfunction, systemic inflammation, and platelet activation. The investigators will test our central hypothesis by carrying out these specific aims: (1) to determine whether eIMPACT reduces the excess CVD risk of depressed patients (primary outcome: endothelial dysfunction; exploratory outcome: incident CVD events) and (2) to examine candidate mechanisms underlying the effect of eIMPACT on CVD risk (secondary outcomes: depressive symptoms, autonomic dysfunction, systemic inflammation, and platelet activation). A positive trial would generate the mechanistic rationale, efficacy evidence, and effect size estimates needed to justify and design a multisite, event-driven, phase III trial to confirm eIMPACT's efficacy in reducing CVD risk. Demonstrating that depression treatment reduces CVD risk, the primary expected outcome of this line of research, would have a substantial positive impact. It would identify a novel target (depression) for CVD prevention efforts, and it would equip providers with a new disseminable and scalable tool (eIMPACT) to simultaneously treat depression and manage the CVD risk of a large cohort of high-risk patients. Collectively, these changes to clinical practice should translate into reduced CVD morbidity, mortality, and costs.

ELIGIBILITY:
Inclusion Criteria:

* Primary care patients
* Age ≥ 50 years
* Current depressive disorder
* Elevated cardiovascular disease risk

Exclusion Criteria:

* History of clinical cardiovascular disease
* Presence of the following chronic disorders: HIV/AIDS, chronic kidney disease, systemic inflammatory disease, or past-year cancer
* History of bipolar disorder or psychosis
* Continuous (e.g., daily) treatment for a systemic inflammatory condition (e.g., rheumatoid arthritis, lupus, Crohn's disease, and ulcerative colitis) in the past 3 months. Nonsteroidal anti-inflammatory drug (NSAID) use is allowed, given its high prevalence in the target population.
* Current use of anticoagulants (Aspirin and cholesterol and blood pressure medications are allowed)
* Acute risk of suicide
* Severe cognitive impairment
* Current pregnancy
* Ongoing depression treatment with a psychiatrist outside of the Eskenazi Health/Midtown system (ongoing depression treatment with a Eskenazi Health/Midtown psychiatrist is allowed, as we will be able to collaborate and coordinate depression care)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse C Stewart, Ph.D., Principal Investigator — Indiana University-Purdue University Indianapolis (IUPUI)
Locations (1):
- IUPUI Department of Psychology, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Williams MK, Shell AL, Wu W, MacDonald KL, Callahan CM, Nurnberger JI Jr, Crawford CA, Schuiling MD, Stewart JC. Longer-term effects of modernized collaborative care for depression on multiple mental health factors (eIMPACT): A randomized controlled trial. J Affect Disord. 2026 Jan 1;392:120272. doi: 10.1016/j.jad.2025.120272. Epub 2025 Sep 8. PMID 40930184
- [Derived] Schuiling MD, Wu W, Polanka BM, Shell AL, Williams MK, Crawford CA, MacDonald KL, Nurnberger JI Jr, Callahan CM, Stewart JC. Effect of depression treatment on subjective sleep components among primary care patients: Data from the eIMPACT trial. J Mood Anxiety Disord. 2025 Jun 3;11:100132. doi: 10.1016/j.xjmad.2025.100132. eCollection 2025 Sep. PMID 40822596
- [Derived] Schuiling MD, Shell AL, Callahan CM, Nurnberger JI Jr, MacDonald KL, Considine RV, Wu W, Hirsh AT, Crawford CA, Williams MK, Lipuma TC, Gupta SK, Kovacs RJ, Rollman BL, Stewart JC. Effect of depression treatment on health behaviors and cardiovascular risk factors in primary care patients with depression and elevated cardiovascular risk: data from the eIMPACT trial. Psychol Med. 2024 Sep 10:1-14. doi: 10.1017/S0033291724001429. Online ahead of print. PMID 39252547
- [Derived] Crawford CA, Williams MK, Shell AL, MacDonald KL, Considine RV, Wu W, Rand KL, Stewart JC. Effect of modernized collaborative care for depression on brain-derived neurotrophic factor (BDNF) and depressive symptom clusters: Data from the eIMPACT trial. Psychiatry Res. 2023 Dec;330:115581. doi: 10.1016/j.psychres.2023.115581. Epub 2023 Oct 30. PMID 37931480
- [Derived] Stewart JC, Patel JS, Polanka BM, Gao S, Nurnberger JI, MacDonald KL, Gupta SK, Considine RV, Kovacs RJ, Vrany EA, Berntson J, Hsueh L, Shell AL, Rollman BL, Callahan CM. Effect of modernized collaborative care for depression on depressive symptoms and cardiovascular disease risk biomarkers: eIMPACT randomized controlled trial. Brain Behav Immun. 2023 Aug;112:18-28. doi: 10.1016/j.bbi.2023.05.007. Epub 2023 May 18. PMID 37209779
- [Derived] Shell AL, Gonzenbach V, Sawhney M, Crawford CA, Stewart JC. Associations between affective factors and high-frequency heart rate variability in primary care patients with depression. J Psychosom Res. 2022 Oct;161:110992. doi: 10.1016/j.jpsychores.2022.110992. Epub 2022 Jul 22. PMID 35917659

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | eIMPACT | Usual Care
Started | 107 | 109
Completed | 99 | 100
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | eIMPACT | Usual Care | Total
Number analyzed (Participants) | 107 | 109 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (6.0) | 58.9 (5.4) | 58.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 86 | 169
  Male | 24 | 23 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 102 | 104 | 206
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 56 | 51 | 107
  White | 45 | 52 | 97
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 107 | 109 | 216
Brachial Artery Flow-Mediated Dilation [Mean (Standard Deviation); unit: % increase in brachial diameter] — Brachial FMD was measured per consensus guidelines using a GE LOGIQe high-resolution ultrasound with a 15-MHz vascular transducer. After a 10-minute supine rest period, a BP cuff was placed on the forearm and inflated to 250 mmHg for five minutes. Brachial diameter was measured at pre-inflation and 60- and 90-seconds post-deflation using AccessPoint 2011 software (version 8.2). FMD was computed the maximum % increase in brachial diameter at 60- or 90-seconds post-deflation.
  % increase in brachial diameter | 2.59 (2.16) | 2.85 (2.45) | 2.72 (2.31)
Depressive Symptoms [Mean (Standard Deviation); unit: Score on a scale] — Participants completed the reliable and valid Hopkins Symptom Checklist-20 (SCL-20) to assess depressive symptoms. Total scores (mean of items responses, range: 0-4) were computed, with higher scores indicating greater depressive symptoms.
  Score on a scale | 1.86 (0.76) | 1.96 (0.68) | 1.91 (0.72)
High-Frequency Heart Rate Variability (HF HRV) [Mean (Standard Deviation); unit: ln of ms^2/Hz] — HF HRV estimates were derived by spectral analysis (bandwidth: 0.15-0.40 Hz) from 1-minute epochs of electrocardiographic data obtained during the last 5 min of the 10-minute supine rest period using MindWare Technologies HRV analysis software (version 3.1.2). Mean HF HRV was computed as the average of the five estimates. To control for respiration rate, participants completed a paced-breathing computer task set to 12 breaths/minute.
  ln of ms^2/Hz | 5.29 (1.72) | 5.15 (1.66) | 5.22 (1.71)
Interleukin-6 (IL-6) [Mean (Standard Deviation); unit: log10 of pg/ml] — Fasting blood samples obtained by research nurses were collected in EDTA tubes and centrifuged within 20 min. Plasma aliquots were frozen at -80 °C until the time of assay at the Indiana University Center for Diabetes and Metabolic Diseases Translation Core. Using enzyme-linked immunosorbent assay kits according to the manufacturer's instructions, we measured levels of IL-6.
  log10 of pg/ml | 0.71 (0.28) | 0.75 (0.27) | 0.73 (0.27)
High-Sensitivity C-Reactive Protein (hsCRP) [Mean (Standard Deviation); unit: log10 of mg/l] — Fasting blood samples obtained by research nurses were collected in EDTA tubes and centrifuged within 20 min. Plasma aliquots were frozen at -80 °C until the time of assay at the Indiana University Center for Diabetes and Metabolic Diseases Translation Core. Using enzyme-linked immunosorbent assay kits according to the manufacturer's instructions, we measured levels of hsCRP.
  log10 of mg/l | 0.67 (0.40) | 0.71 (0.40) | 0.69 (0.40)
β-thromboglobulin [Mean (Standard Deviation); unit: ng/ml] — Fasting blood samples obtained by research nurses were collected in EDTA tubes and centrifuged within 20 min. Plasma aliquots were frozen at -80 °C until the time of assay at the Indiana University Center for Diabetes and Metabolic Diseases Translation Core. Using enzyme-linked immunosorbent assay kits according to the manufacturer's instructions, we measured levels of β-thromboglobulin.
  ng/ml | 194 (118) | 213 (108) | 204 (113)
Platelet Factor 4 (PF4) [Mean (Standard Deviation); unit: ng/ml] — Fasting blood samples obtained by research nurses were collected in EDTA tubes and centrifuged within 20 min. Plasma aliquots were frozen at -80 °C until the time of assay at the Indiana University Center for Diabetes and Metabolic Diseases Translation Core. Using enzyme-linked immunosorbent assay kits according to the manufacturer's instructions, we measured levels of PF4.
  ng/ml | 4038 (2047) | 4290 (2133) | 4165 (2094)

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Flow-Mediated Dilation (FMD) at 12 Months
Description: Brachial FMD was measured per consensus guidelines using a GE LOGIQe high-resolution ultrasound with a 15-MHz vascular transducer. After a 10-minute supine rest period, a BP cuff was placed on the forearm and inflated to 250 mmHg for five minutes. Brachial diameter was measured at pre-inflation and 60- and 90-seconds post-deflation using AccessPoint 2011 software (version 8.2). FMD was computed the maximum % increase in brachial diameter at 60- or 90-seconds post-deflation.
Time Frame: 12 months
Population: 195 of 216 randomized participants had post-treatment brachial FMD data. Because multiple imputation was employed, all 216 randomized participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: % increase in brachial diameter
Arm/Group | eIMPACT | Usual Care
Number analyzed (Participants) | 107 | 109
% increase in brachial diameter | 2.28 (2.04) | 2.44 (2.29)
Statistical Analysis 1: Comparison: eIMPACT vs Usual Care; Test type: Superiority; p = 0.60, ANCOVA; ANCOVA models adjusted for the stratification variables of age group and sex

2. Secondary Outcome: Depressive Symptoms at 12 Months
Description: Participants completed the reliable and valid Hopkins Symptom Checklist-20 (SCL-20) to assess depressive symptoms. Total scores (mean of items responses, range: 0-4) were computed, with higher scores indicating greater depressive symptoms.
Time Frame: 12 months
Population: 200 of 216 randomized participants had post-treatment SCL-20 data. Because multiple imputation was employed, all 216 randomized participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | eIMPACT | Usual Care
Number analyzed (Participants) | 107 | 109
Score on a scale | 1.12 (0.80) | 1.65 (0.83)
Statistical Analysis 1: Comparison: eIMPACT vs Usual Care; Test type: Superiority; p < 0.01, ANCOVA; ANCOVA models adjusted for the stratification variables of age group and sex

3. Secondary Outcome: High-Frequency Heart Rate Variability (HF HRV) at 12 Months
Description: HF HRV estimates were derived by spectral analysis (bandwidth: 0.15-0.40 Hz) from 1-minute epochs of electrocardiographic data obtained during the last 5 min of the 10-minute supine rest period using MindWare Technologies HRV analysis software (version 3.1.2). Mean HF HRV was computed as the average of the five estimates. To control for respiration rate, participants completed a paced-breathing computer task set to 12 breaths/minute.
Time Frame: 12 months
Population: 190 of 216 randomized participants had post-treatment SCL-20 data. Because multiple imputation was employed, all 216 randomized participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: ln of ms^2/Hz
Arm/Group | eIMPACT | Usual Care
Number analyzed (Participants) | 107 | 109
ln of ms^2/Hz | 5.39 (1.85) | 5.35 (1.78)
Statistical Analysis 1: Comparison: eIMPACT vs Usual Care; Test type: Superiority; p = 0.81, ANCOVA; ANCOVA models adjusted for the stratification variables of age group and sex

4. Secondary Outcome: Interleukin-6 (IL-6) at 12 Months
Description: Fasting blood samples obtained by research nurses were collected in EDTA tubes and centrifuged within 20 min. Plasma aliquots were frozen at -80 °C until the time of assay at the Indiana University Center for Diabetes and Metabolic Diseases Translation Core. Using enzyme-linked immunosorbent assay kits according to the manufacturer's instructions, we measured levels of IL-6.
Time Frame: 12 months
Population: 195 of 216 randomized participants had post-treatment SCL-20 data. Because multiple imputation was employed, all 216 randomized participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: log10 of pg/ml
Arm/Group | eIMPACT | Usual Care
Number analyzed (Participants) | 107 | 109
log10 of pg/ml | 0.73 (0.26) | 0.77 (0.27)
Statistical Analysis 1: Comparison: eIMPACT vs Usual Care; Test type: Superiority; p = 0.20, ANCOVA; ANCOVA models adjusted for the stratification variables of age group and sex

5. Secondary Outcome: High-Sensitivity C-Reactive Protein (hsCRP) at 12 Months
Description: Fasting blood samples obtained by research nurses were collected in EDTA tubes and centrifuged within 20 min. Plasma aliquots were frozen at -80 °C until the time of assay at the Indiana University Center for Diabetes and Metabolic Diseases Translation Core. Using enzyme-linked immunosorbent assay kits according to the manufacturer's instructions, we measured levels of hsCRP.
Time Frame: 12 months
Population: 196 of 216 randomized participants had post-treatment SCL-20 data. Because multiple imputation was employed, all 216 randomized participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: log10 of mg/l
Arm/Group | eIMPACT | Usual Care
Number analyzed (Participants) | 107 | 109
log10 of mg/l | 0.65 (0.40) | 0.74 (0.41)
Statistical Analysis 1: Comparison: eIMPACT vs Usual Care; Test type: Superiority; p = 0.09, ANCOVA; ANCOVA models adjusted for the stratification variables of age group and sex

6. Secondary Outcome: β-thromboglobulin at 12 Months
Description: Fasting blood samples obtained by research nurses were collected in EDTA tubes and centrifuged within 20 min. Plasma aliquots were frozen at -80 °C until the time of assay at the Indiana University Center for Diabetes and Metabolic Diseases Translation Core. Using enzyme-linked immunosorbent assay kits according to the manufacturer's instructions, we measured levels of β-thromboglobulin.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | eIMPACT | Usual Care
Number analyzed (Participants) | 107 | 109
ng/ml | 185 (125) | 205 (118)
Statistical Analysis 1: Comparison: eIMPACT vs Usual Care; Test type: Superiority; p = 0.23, ANCOVA; ANCOVA models adjusted for the stratification variables of age group and sex

7. Secondary Outcome: Platelet Factor 4 (PF4) at 12 Months
Description: Fasting blood samples obtained by research nurses were collected in EDTA tubes and centrifuged within 20 min. Plasma aliquots were frozen at -80 °C until the time of assay at the Indiana University Center for Diabetes and Metabolic Diseases Translation Core. Using enzyme-linked immunosorbent assay kits according to the manufacturer's instructions, we measured levels of PF4.
Time Frame: 12 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | eIMPACT | Usual Care
Number analyzed (Participants) | 107 | 109
ng/ml | 3842 (2011) | 4351 (2341)
Statistical Analysis 1: Comparison: eIMPACT vs Usual Care; Test type: Superiority; p = 0.09, ANCOVA; ANCOVA models adjusted for the stratification variables of age group and sex

ADVERSE EVENTS:
Time Frame: For each participant, adverse event monitoring occurred from each participant's randomization date until 9/1/20 (the date of the last EHR for all randomized participants). Thus, the adverse event monitoring period varied across participants but averaged 3.5 years.
Description: Potential adverse events are identified by conducting EHR searches every 6 months and by reviewing self-report adverse event questionnaires from mid-treatment, post-treatment, and the annual follow-up calls. We investigate, rate, and write up all events plausibly related to depression, depression treatment, suicidal ideation, or any study procedures. We adjudicate all deaths. For all other captured events, we provide counts and will investigate further if there is evidence of group imbalance.
Arm/Group | eIMPACT | Usual Care
All-Cause Mortality (participants affected / at risk) | 5/107 | 8/109
Serious Adverse Events (participants affected / at risk) | 5/107 | 4/109
Other Adverse Events (participants affected / at risk) | 3/107 | 1/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | eIMPACT (N=107) | Usual Care (N=109)
Hospitalization for depression/suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1)
Emergency department visit for depression/suicidal ideation (Psychiatric disorders) | 2 (3) | 1 (1)
Suspected drug overdose (Psychiatric disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Endocrine disorders) | 0 (0) | 1 (1)
Study procedures, including depression treatment (Psychiatric disorders) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | eIMPACT (N=107) | Usual Care (N=109)
Passive suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Diarrhea following study-initiated suicidal ideation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Petechiae on hand/wrist due to blood pressure cuff inflation during brachial FMD assessment (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT02458690/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT02458690/ICF_001.pdf